CLINICAL TRIAL: NCT05375448
Title: Effects of Neurodynamics of Pain and Function in Patients With Knee Osteoarthrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEU-025
Record Dates: First submitted 2022-05-11; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will perform an active femoral nerve mobilisation technique. The treatment will be performed at home.
  Patients will receive a video model to perform the exercise during the 8 weeks of treatment. The treatment should be performed 10 repetitions twice a day, with one set recommended in the morning and one in the evening.
  The treatment will be monitored by telephone and if there are any doubts, the session will be carried out together with the patient.
  Interventions: Other: Neural mobilisation

INTERVENTIONS:
Other: Neural mobilisation — Participants will perform an active femoral nerve mobilisation technique. The treatment will be performed at home.
  Patients will receive a video model to perform the exercise during the 8 weeks of treatment. The treatment should be performed 10 repetitions twice a day, with one set recommended in the morning and one in the evening.
  The treatment will be monitored by telephone and if there are any doubts, the session will be carried out together with the patient.

SUMMARY:
Osteoarthritis is defined as a degenerative joint disease characterised by a decrease in joint space due to cartilage loss and the presence of subchondral sclerosis and osteophytes. It is the most common joint disease and is expected to become the fourth leading cause of disability worldwide by 2020. The knee is the joint most affected by osteoarthritis.

The prevalence of osteoarthritis of the knee has been increasing in recent years. The main risk factors are female sex, although in recent years there has been a greater relative increase in men, comorbidity, age, mechanical stress and obesity, the latter being of great importance in the progression and development of osteoarthritis.

There are two types of osteoarthritis of the knee, primary (idiopathic) and secondary (previous causal alteration). This disease causes pain and disability, so that these patients have difficulty walking, standing, sitting, climbing and descending stairs, resulting in decreased function and negatively impacting the performance of activities of daily living.

The Kellgren and Lawrence scale, which marks the degree of involvement of osteoarthritis by the level of joint destruction based on radiography, is a validated method that gives us IV degrees of the disease, with grade I being the mildest and IV the most severe.

Pain in this syndrome is a multifactorial phenomenon involving neurophysiological, structural and psychosocial factors (10). In relation to neurophysiological factors, it has been shown that inflammatory mediators in somatic structures alter afferent sensory inputs and induce plastic changes in the nervous system, which can lead to central sensitisation (CS).

Sensitisation is defined as an increased response to a painful stimulus by increasing the signal in the central nervous system, either by decreasing the activation of descending inhibitory pain systems or by increasing the pain signal.

MRI studies have also shown that patients with osteoarthritis of the knee have a lower degree of disengagement and increased pain vigilance, associated with abnormal activity in different areas of the brain such as the cingulate cortex, insula, amygdala, prefrontal areas and nucleus accubens.

Currently, conservative treatment of osteoarthritis of the knee is aimed at reducing pain, increasing function and reducing joint damage by means of pharmacological and non-pharmacological therapies. Pharmacological treatment is based primarily on paracetamol and non-steroidal anti-inflammatory drugs (NSAIDs), but these drugs are associated with adverse effects, especially at older ages. As for non-pharmacological therapy, we mainly find exercise-based treatment and manual therapy-based treatment, both showing improvements in pain and function of patients and showing better results in combination.

Neural mobilisation consists of sliding the nerves, seeking to restore the dynamic balance between the nerve and associated tissues, thus increasing vascularisation, decreasing neural pressure and eliminating harmful fluids. There are studies showing how this technique improves range of motion and knee pain, but more literature on this technique is needed.Our hypothesis is that femoral nerve mobilisation can have a positive effect on function and a decrease in pain in patients with grades I-II osteoarthritis of the knee, with neurodynamics being a possible treatment for these patients.

Aims:

To determine the effectiveness of treatment with femoral nerve neurodynamics in patients with osteoarthritis of the knee. Assessing the decrease in pain and increase in function by means of pain intensity, pressure pain thresholds, temporal assessment, pain modulation, KOOS, SF-12 and CSI questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis, grade I and II, of the Kellgren Lawrence scale.
* Knee pain diagnosed as osteoarthritis of the knee using the American College of Rheumatology criteria.

Exclusion Criteria:

* Disorders, syndromes or diseases that may cause myofascial or neuropathic pain in the lower limbs, such as lumbar radiculopathy, meralgia paraesthetica or saphenous nerve entrapment.
* Chronic diseases that may be considered perpetuating factors such as fibromyalgia
* Corticosteroid or local anaesthetic injections during the year prior to the patient's participation in the study or during follow-up.
* Consumption of oral analgesics on a constant basis and 24 h before the measurements.
* Ingesting substances of abuse that may interfere during treatment such as alcohol and drugs.
* Cognitive deficit manifested in the clinical history (Alzheimer, dementia) or measured by the Mini-Cognitive Examination

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale | 12 months
  The Numerical Rating Scale (NRS) will be used with 11 intervals with a score of 0-10, where 0 would correspond to no pain and 10 to the worst pain imaginab
threshold pain | 12 months
  To measure pressure pain thresholds, we use an algometer with a surface area of 1 cm2 , applying it perpendicularly to the skin at a speed of 1 kg/cm2/s until the patient indicates that the first sensation of pain appears, at which point the pressure applied stops.
SF-12 | 12 months
  It is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
  The SF-12 is a shortened version of the SF-36.
KOOS questionnaire | 12 months
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a questionnaire designed to assess short and long-term patient-relevant outcomes following knee injury. The KOOS is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. The KOOS meets basic criteria of outcome measures and can be used to evaluate the course of knee injury and treatment outcome. KOOS is patient-administered, the format is user-friendly and it takes about 10 minutes to fill out

SECONDARY OUTCOMES:
Pain modulation | 12 months
  We combine temporary assessment and a sphygmomanometer on the contralateral arm of the knee with osteoarthritis. It is inflated at a rate of 20 mm Hg/s until the first sensation of pain and held for 30 seconds. The sphygmomanometer shall be inflated or deflated until a pain intensity of 3/10 on the numerical pain rating scale is achieved. The temporary assessment shall then be repeated with inflation of the sphygmomanometer
Temporal variation of pain | 12 months
  pressure pain thresholds shall be measured. Subsequently, 10 consecutive pulses shall be made at the same locations to elicit the temporary assessment, increasing the pressure by 2 kg/s and maintained for 1 second (followed by 1 second of rest) at each pulse. The intensity of pain at the 1st, 5th and 10th pulse shall be assessed by means of a numerical pain scale (0 being no pain and 10 being the maximum pain imaginable).

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Juan-Carlos Zuil-Escobar, Alcorcón
  - CEU-San Pablo Universtiy, Madrid